CLINICAL TRIAL: NCT04984122
Title: Influence of General and Local Anesthesia on Postoperative Pain After Loop Electrosurgical Excision Procedure: A Randomized Trial
Brief Title: Anesthesia on Postoperative Pain After Loop Electrosurgical Excision Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Medical Doctor - Professor, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUGLA-5
Record Dates: First submitted 2021-07-25; First posted 2021-07-30 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Procedure, Gynecologic Surgical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): GA group intravenous 2-3 μ/kg fentanyl followed by 2 mg/kg propofol. were administered for anesthesia induction. After a laryngeal mask insertion anesthesia was maintained by inhalation of sevoflurane in an oxygen (60%) and nitrous oxide (40%) mixture to maintain a minimal alveolar concentration (MAC) of 0.8%-1.3%.
  Interventions: Procedure: LEEP
- Study (Other): In the LA group, after positioning of the patient, 50 mg of lidocaine spray (5 pumps, 10 mg in each pump) were applied to the ectocervix, then 2 mL bupivacaine hydrochloride was injected submucosally using a 27-gauge needle tip at the 3, 6, 9, and 12 o'clock locations in the ectocervix.
  Interventions: Procedure: LEEP

INTERVENTIONS:
Procedure: LEEP — According to the size of the cervix, a loop electrode size was selected. The electrical power for the loop electrode was set to 50 W cut and 45 W coagulation in blended mode. LEEP was performed by carefully passing the loop around the transformation zone from 12 o'clock to 6 o'clock. An additional top-hat excision was performed in patients with a lesion deep in the cervical canal. After completion of the excision, hemostasis was exclusively obtained using the ball electrode in spray coagulation mode. No suturing or other methods were used for hemostasis.

SUMMARY:
The loop electrosurgical excision procedure (LEEP) is a modified cervical conization that is performed with an electrosurgical loop. It may be performed under local anesthesia (LA) or under general anesthesia (GA), and practice patterns differ widely. In some countries, specific guidelines for the choice of anesthesia during LEEP are provided, whereas, in other countries, the choice of anesthesia is not specified. LEEP under LA is more economical, obviating the need for anesthesia staff, equipment, and operating room fees. However, LEEP under LA may be more difficult to perform, may be more difficult to learn, may lead to inferior surgical results, and may result in more pain and patient dissatisfaction. This study aimed to compare loop electrosurgical excision procedures under local anesthesia vs general anesthesia regarding patients' satisfaction, histopathologic results, and short-term morbidity

ELIGIBILITY:
Inclusion Criteria:

Patients were > 21 years old; were not pregnant

The patient had one of the following indications for LEEP:

1. histologyproven, persistent, low-grade squamous intraepithelial lesion (LGSIL);
2. a histology-proven high-grade squamous intraepithelial lesion (HGSIL);
3. discrepancies between cytological reports and colposcopic impressions;
4. investigation for unsatisfactory colposcopy;
5. microinvasion or adenocarcinoma in situ on cervical punch biopsy.

Exclusion Criteria:

Patients with cervical or vaginal infection; Patients with an abnormal menstrual cycle; who were taking anticoagulants, Patients with a coagulation defect Patients with mental incapacity Patients with previous hysterectomy with removal of the cervix Patients with a history of cervical cancer.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
visual analog scale 1 | up to 1 hour after the procedure
  VAS score ( 0 cm = no pain, 10 cm = worst pain imaginable) reported for the pain felt at 1 hour after procedure.

SECONDARY OUTCOMES:
visual analog scale 2 | up to 2 hour after the procedure
  VAS score ( 0 cm = no pain, 10 cm = worst pain imaginable) reported for the pain felt at 2 hours after LEEP

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kemal Gungorduk, Muğla
  - Mugla Sıtkı Kocman University Education and Research Hospital, Muğla

IPD SHARING:
Plan to Share IPD: Undecided